CLINICAL TRIAL: NCT02314780
Title: Pilot Trial: The Effects of Intravenous Heme Arginate on HO-1 Expression and Oxidative Stress in the Human Heart
Brief Title: The Effects of Intravenous Heme Arginate on Heme Oxygenase-1 Expression (HO-1) and Oxidative Stress in the Human Heart
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Martin Andreas, M.D. (Other)
Collaborators: National Bank of Austria (Other Government); Orphan Medical (Industry)
Responsible Party: Sponsor-Investigator, Martin Andreas, M.D., M.D., PhD, Medical University of Vienna
Organization: Medical University of Vienna (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HO-1 in the Heart; 2013-000887-27 (EudraCT Number)
Record Dates: First submitted 2014-12-08; First posted 2014-12-11 (Estimated); Results first posted 2021-02-15 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2021-01

CONDITIONS: Myocardial Ischemia
Keywords: carboxyhemoglobin; neutrophil; reactive oxygen species; reperfusion injury
MeSH Terms: conditions — Myocardial Ischemia; Reperfusion Injury | interventions — heme arginate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Heme arginate (high dose) (Experimental): 24 hours prior to the planned surgical aortic valve replacement, heme arginate at a dose of 3 mg/kg diluted to 110ml with 0.9% sodium chloride was administered at a single intravenous infusion using an infusion pump.
  Interventions: Drug: Heme arginate 3mg/kg
- Heme arginate (low dose) (Experimental): 24 hours prior to the planned surgical aortic valve replacement, heme arginate at a dose of 1 mg/kg diluted to 110ml with 0.9% sodium chloride was administered at a single intravenous infusion using an infusion pump.
  Interventions: Drug: Heme arginate 1mg/kg
- Placebo (Placebo Comparator): 24 hours prior to the planned surgical aortic valve replacement, subjects received a single intravenous infusion of an equivalent volume of 0.9% sodium chloride solution.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Heme arginate 3mg/kg
  Other Names: Normosang
  Arms: Heme arginate (high dose)
Drug: Heme arginate 1mg/kg
  Other Names: Normosang
  Arms: Heme arginate (low dose)
Drug: Placebo
  Other Names: 0.9% sodium chloride solution
  Arms: Placebo

SUMMARY:
Ischemia reperfusion injury may be attenuated by HO-1 induction. Our previous data confirmed strong HO-1 induction in peripheral blood cells following heme arginate infusion in healthy humans. Furthermore, we could demonstrate the amelioration of experimental ischemia reperfusion injury in the calf musculature by heme arginate in healthy subjects as measured by functional MRI.

Therefore, we propose that HO-1 induction in the human heart may be a suitable target to mitigate cardiac ischemia-reperfusion injury.

The HO-1 induction will be assessed in a clinical trial by myocardial biopsy prior to and after aortic cross-clamping in subjects with or without preceding heme arginate treatment in two different dosages. The HO-1 expression will also be measured in the clinical trials in peripheral blood mononuclear cells. As additional outcome, levels of myoglobin, creatine-kinase and troponin T and reactive oxygen species will be measured in plasma according to standard laboratory procedures.

ELIGIBILITY:
Inclusion criteria:

* Signed informed consent
* Men and women aged between 40 and 85 years (inclusive)
* Body mass index < 35 kg/m2
* Ability to communicate well with the investigator in the local language and to understand and comply with the requirements of the study

Exclusion criteria (any of the following):

* Known hypersensitivity to the study drug or any excipients of the drug formulation
* Treatment with another investigational drug within 3 weeks prior to screening
* History or clinical evidence of any disease and/or existence of any surgical or medical condition, which might interfere with the absorption, distribution, metabolism or excretion of the study drug
* Severe renal failure (glomerula filtration rate < 30 ml/min)
* Moderately or severe impaired left ventricular function (ejection fraction < 40%)
* Moderately or severe impaired right ventricular function
* Systolic pulmonary pressure > 45 mmHg
* Acute or recent (<7 days) myocardial infarction
* Child bearing potential

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2015-03-29 (Actual); Primary Completion 2017-06-13 (Actual); Study Completion 2017-06-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alfred Kocher, M.D., Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

REFERENCES:
- [Derived] Andreas M, Oeser C, Kainz FM, Shabanian S, Aref T, Bilban M, Messner B, Heidtmann J, Laufer G, Kocher A, Wolzt M. Intravenous Heme Arginate Induces HO-1 (Heme Oxygenase-1) in the Human Heart. Arterioscler Thromb Vasc Biol. 2018 Nov;38(11):2755-2762. doi: 10.1161/ATVBAHA.118.311832. PMID 30354231

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients who were scheduled for elective surgical aortic valve replacement were assessed for eligibility after hospitalization at the Medical University of Vienna.
Pre-assignment Details: A total of 31 patients signed the informed consent to participate in the study. Of them, 27 patients were assigned to a group and 4 patients (3 patients for organizational reasons and 1 patient for other reasons) were excluded from the study prior to assignment to a group.
Period: Overall Study
Arm/Group | Heme Arginate (High Dose) | Heme Arginate (Low Dose) | Placebo
Started | 9 | 10 | 8
Completed | 9 | 7 | 8
Not Completed | 0 | 3 | 0
Not completed — organizational reasons | 0 | 2 | 0
Not completed — Adverse Event | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Heme Arginate (High Dose) | Heme Arginate (Low Dose) | Placebo | Total
Number analyzed (Participants) | 9 | 10 | 8 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 3 | 6
  >=65 years | 7 | 9 | 5 | 21
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 5 | 16
  Male | 3 | 5 | 3 | 11
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Austria | 9 | 10 | 8 | 27

OUTCOME MEASURES:

1. Primary Outcome: Heme Oxygenase-1 (HO-1) Messenger Ribonucleic Acid (mRNA) Levels (Atrial Tissue)
Description: The right atrial appendage was clamped and cut for cannulation before cardiopulmonary bypass. The tissue samples were snap-frozen in the operating theater after sampling.
Time Frame: intraoperative
Measure: Mean (Standard Deviation); unit: arbitrary units
Arm/Group | Heme Arginate (High Dose) | Heme Arginate (Low Dose) | Placebo
Number analyzed (Participants) | 9 | 7 | 8
arbitrary units | 392.7 (195.7) | 229.8 (173.1) | 10.8 (8.8)
Statistical Analysis 1: Comparison: Heme Arginate (High Dose) vs Heme Arginate (Low Dose) vs Placebo; Test type: Other; p = 0.001, ANOVA

2. Primary Outcome: Myocardial HO-1 mRNA Levels (Ventricular Tissue Before Aortic Cross-clamping)
Description: A small biopsy was taken from the right ventricular free wall directly before aortic cross-clamping. The tissue samples were snap-frozen in the operating theater after sampling.
Time Frame: intraoperative
Measure: Mean (Standard Deviation); unit: arbitrary units
Arm/Group | Heme Arginate (High Dose) | Heme Arginate (Low Dose) | Placebo
Number analyzed (Participants) | 9 | 7 | 8
arbitrary units | 203.6 (148.7) | 88.6 (49.1) | 7.9 (5.0)
Statistical Analysis 1: Comparison: Heme Arginate (High Dose) vs Heme Arginate (Low Dose) vs Placebo; Test type: Other; p = 0.002, ANOVA

3. Primary Outcome: Myocardial HO-1 mRNA Levels (Ventricular Tissue After Aortic Cross-clamping)
Description: A small biopsy was taken from the right ventricular free wall after aortic clamp release before weaning from cardiopulmonary bypass. The tissue samples were snap-frozen in the operating theater after sampling.
Time Frame: intraoperative
Measure: Mean (Standard Deviation); unit: arbitrary units
Arm/Group | Heme Arginate (High Dose) | Heme Arginate (Low Dose) | Placebo
Number analyzed (Participants) | 9 | 7 | 8
arbitrary units | 219.4 (162.8) | 108.1 (73.2) | 8.3 (5.4)
Statistical Analysis 1: Comparison: Heme Arginate (High Dose) vs Heme Arginate (Low Dose) vs Placebo; Test type: Other; p = 0.002, ANOVA

4. Primary Outcome: Myocardial HO-1 Protein Concentrations (Atrial Tissue)
Description: The right atrial appendage was clamped and cut for cannulation before cardiopulmonary bypass.The tissue samples were snap-frozen. Western blot analysis was performed. The amount of HO-1 protein (quantified as pixels under the curve) was evaluated.
Time Frame: intraoperative
Measure: Mean (Standard Deviation); unit: pixels under the curve
Arm/Group | Heme Arginate (High Dose) | Heme Arginate (Low Dose) | Placebo
Number analyzed (Participants) | 9 | 7 | 8
pixels under the curve | 29022 (8583) | 28585 (10692) | 8401 (3889)
Statistical Analysis 1: Comparison: Heme Arginate (High Dose) vs Heme Arginate (Low Dose) vs Placebo; Test type: Other; p < 0.001, ANOVA

5. Primary Outcome: Myocardial HO-1 Protein Concentrations (Ventricular Tissue Before Aortic Cross-clamping)
Description: A small biopsy was taken from the right ventricular free wall directly before aortic cross-clamping. The tissue samples were snap-frozen. Western blot analysis was performed. The amount of HO-1 protein (quantified as pixels under the curve) was evaluated.
Time Frame: intraoperative
Measure: Mean (Standard Deviation); unit: pixels under the curve
Arm/Group | Heme Arginate (High Dose) | Heme Arginate (Low Dose) | Placebo
Number analyzed (Participants) | 9 | 7 | 8
pixels under the curve | 13752 (8069) | 10534 (4686) | 6842 (4343)
Statistical Analysis 1: Comparison: Heme Arginate (High Dose) vs Heme Arginate (Low Dose) vs Placebo; Test type: Other; p = 0.138, ANOVA

6. Primary Outcome: Myocardial HO-1 Protein Concentrations (Ventricular Tissue After Aortic Cross-clamping)
Description: A small biopsy was taken from the right ventricular free wall after aortic clamp release before weaning from cardiopulmonary bypass. The tissue samples were snap-frozen in the operating theater after sampling. Western blot analysis was performed. The amount of HO-1 protein (quantified as pixels under the curve) was evaluated.
Time Frame: intraoperative
Measure: Mean (Standard Deviation); unit: pixels under the curve
Arm/Group | Heme Arginate (High Dose) | Heme Arginate (Low Dose) | Placebo
Number analyzed (Participants) | 9 | 7 | 8
pixels under the curve | 17062 (18164) | 11277 (3918) | 12037 (10962)
Statistical Analysis 1: Comparison: Heme Arginate (High Dose) vs Heme Arginate (Low Dose) vs Placebo; Test type: Other; p = 0.696, ANOVA

ADVERSE EVENTS:
Time Frame: Adverse events occuring within 96 hours after the administration of heme arginate/sodium chloride solution were reported.
Arm/Group | Heme Arginate (High Dose) | Heme Arginate (Low Dose) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/10 | 0/8
Serious Adverse Events (participants affected / at risk) | 2/9 | 0/10 | 1/8
Other Adverse Events (participants affected / at risk) | 1/9 | 5/10 | 4/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Heme Arginate (High Dose) (N=9) | Heme Arginate (Low Dose) (N=10) | Placebo (N=8)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Coronary artery compression (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Heme Arginate (High Dose) (N=9) | Heme Arginate (Low Dose) (N=10) | Placebo (N=8)
Procedural pneumothorax (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Blood culture positive (Investigations) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 3 (3) | 3 (3)
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Acute stress disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Biopsy samples were small and protein concentration could not be measured in every sample. The sample size calculation was based on previous results but is small for a 3-arm randomized controlled trial. Additional surgical procedures might impact the postoperative course of cardiac enzymes and obscure a potential effect in this small group. This study was powered to identify protein expression in the heart but not to evaluate potential therapeutic effects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-05-08): https://cdn.clinicaltrials.gov/large-docs/80/NCT02314780/Prot_SAP_000.pdf